CLINICAL TRIAL: NCT00370435
Title: An Open-label, Single Dose Study to Investigate the Safety, Tolerability and Pharmacokinetics of 90mg of GW274150 in Adult and Elderly RA Subjects.
Brief Title: Study Of 90mg Of GW274150 In Subjects Over 50 Years, Who Have Rheumatoid Arthritis (RA)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 104916
Record Dates: First submitted 2006-08-17; First posted 2006-08-31 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Arthritis, Rheumatoid
Keywords: rheumatoid arthritis; safety; GW274150; pharmacokinetics; tolerability
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — GW 274150

INTERVENTIONS:
Drug: GW274150

SUMMARY:
This is a study of GW274150, an iNOS (inducible nitric oxide synthase) inhibitor to investigate safety, tolerability and pharmacokinetics (PK) in the rheumatoid arthritis (RA) population (greater than 50 years). Safety, tolerability and PK of GW274150 in an adult and elderly population have not yet been determined. Therefore this study is designed to ensure that 90mg GW274150 will be safe and well-tolerated in this adult and elderly RA patient population on methotrexate. The assessments will include pharmacokinetics (PK), liver function tests and creatinine clearance.

This study will provide confidence that a single 90mg dose of GW274150 results in exposure in RA subjects similar to that expected from healthy volunteers and asthmatics.

ELIGIBILITY:
Inclusion criteria:

* No clinically significant disease as determined by history, physical examination and screening investigations.
* RA subjects on methotrexate (7.5mg - 25mg per week)
* Body weight >50 kg for males and >45 kg for females, who are not morbidly obese
* Diagnosis of RA
* Active disease defined as DAS28 = 4.0 and at least one MCP joint with either detectable vascularity or thickness
* Stable doses of DMARDs (Disease-modifying anti-rheumatic drugs, which must include methotrexate and can also include but is not restricted to sulphasalazine and hydroxychloroquine in any combination) for 8 weeks prior to enrolment
* Must be on stable folate supplements
* Subjects using NSAIDs or Cox-2 inhibitors must have been on stable doses for 2 weeks prior to screening
* LFT functions (ALT, AST, ALP) = 1.5 x ULN at screening and which have been stable on at least 2 occasions in the 7 months prior to screening
* Must provide signed and dated written informed consent prior to admission to the study
* Ability to understand and comply with protocol requirements, instructions and protocol-stated restrictions.

Exclusion criteria:

* Past or present disease, which as judged by the investigator, may affect the outcome of this study.
* Clinically significant abnormalities in safety laboratory analysis at screening
* Pregnant or nursing women
* Women of childbearing potential who are unwilling or unable to use an appropriate method of contraception as outlined
* As a result of the medical interview, physical examination or screening investigations, the Physician Responsible considers the subject unfit for the study
* Taking >10mg/day oral glucocorticoids
* Currently receiving anti-rheumatic biological therapy
* Received their final dose of infliximab or adalimumab within 3 months of enrollment
* Received their final dose of etanercept or anakinra within 1 month of enrollment
* Has received an investigational drug or participated in any other NCE research trial within 30 days or 5 half-lives, or twice the duration of the biological effect of any drug (whichever is longer) prior to enrol.ment
* Regularly drinks more than 28 units of alcohol in a week if male, or 21 units per week if female.
* Has a screening QTc value of >430msec (males) or >450msec (females), PR interval outside the range 120 to 200msec or an ECG that is not suitable for QT measurements
* History of liver or renal disease in the 6 months prior to screening
* Current renal insufficiency (subject must have an estimated creatinine clearance less than50mL/min as estimated from the serum creatinine using the Cockroft-Gault formula
* Has donated a unit of blood within the previous month or intends to donate in the month after completing the study
* Has a history or drug or other allergy, which in the opinion of the physician responsible, contraindicates their participation
* History of, or risk factors for, HIV, Hepatitis B and Hepatitis C
* History of drug abuse

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2005-08; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Liver function and creatinine clearance after single 90mg dose of GW274150

SECONDARY OUTCOMES:
clinical laboratory tests assessment of adverse events ECGs vital signs and Pharmacokinetic data of elderly population

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom